CLINICAL TRIAL: NCT00362648
Title: Efficacy, Safety, and Immunogenicity of RotaTeq™ Among Infants in Asia and Africa
Brief Title: Developing World Study for RotaTeq™ (V260-015)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V260-015; 2006_027
Record Dates: First submitted 2006-08-08; First posted 2006-08-10 (Estimated); Results first posted 2010-05-13 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Vomiting; Diarrhea; Fever
MeSH Terms: conditions — Vomiting; Diarrhea; Fever | interventions — RotaTeq; Rotavirus Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): RotaTeq™
  Interventions: Biological: RotaTeq™ - Rotavirus Vaccine, Live, Oral, Pentavalent
- 2 (Placebo Comparator): Placebo
  Interventions: Biological: Comparator: Placebo

INTERVENTIONS:
Biological: RotaTeq™ - Rotavirus Vaccine, Live, Oral, Pentavalent — 2.0 mL oral dose of RotaTeq™. 14 week treatment period
  Other Names: RotaTeq™; V260
  Arms: 1
Biological: Comparator: Placebo — Arm 2: Placebo. 14 week treatment period
  Arms: 2

SUMMARY:
The purpose of the current study is to evaluate whether the vaccine is effective, well-tolerated and immunogenic among infants in developing countries.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 weeks through 12 weeks at Dose 1
* Parent able to understand study procedures and give consent

Exclusion Criteria:

* Clinical evidence of active gastrointestinal disease
* Subjects who are currently or expected to participate in other studies of investigational products during the 6 weeks after receiving the last dose of RotaTeq™/placebo

Ages: 4 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7504 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Gruber JF, Becker-Dreps S, Hudgens MG, Brookhart MA, Thomas JC, Jonsson Funk M. Timing and predictors of severe rotavirus gastroenteritis among unvaccinated infants in low- and middle-income countries. Epidemiol Infect. 2018 Apr;146(6):698-704. doi: 10.1017/S0950268818000626. Epub 2018 Mar 22. PMID 29564996
- [Derived] Gruber JF, Hille DA, Liu GF, Kaplan SS, Nelson M, Goveia MG, Mast TC. Heterogeneity of Rotavirus Vaccine Efficacy Among Infants in Developing Countries. Pediatr Infect Dis J. 2017 Jan;36(1):72-78. doi: 10.1097/INF.0000000000001362. PMID 27755463
- [Derived] Zaman K, Dang DA, Victor JC, Shin S, Yunus M, Dallas MJ, Podder G, Vu DT, Le TP, Luby SP, Le HT, Coia ML, Lewis K, Rivers SB, Sack DA, Schodel F, Steele AD, Neuzil KM, Ciarlet M. Efficacy of pentavalent rotavirus vaccine against severe rotavirus gastroenteritis in infants in developing countries in Asia: a randomised, double-blind, placebo-controlled trial. Lancet. 2010 Aug 21;376(9741):615-23. doi: 10.1016/S0140-6736(10)60755-6. Epub 2010 Aug 6. PMID 20692031
- [Derived] Armah GE, Sow SO, Breiman RF, Dallas MJ, Tapia MD, Feikin DR, Binka FN, Steele AD, Laserson KF, Ansah NA, Levine MM, Lewis K, Coia ML, Attah-Poku M, Ojwando J, Rivers SB, Victor JC, Nyambane G, Hodgson A, Schodel F, Ciarlet M, Neuzil KM. Efficacy of pentavalent rotavirus vaccine against severe rotavirus gastroenteritis in infants in developing countries in sub-Saharan Africa: a randomised, double-blind, placebo-controlled trial. Lancet. 2010 Aug 21;376(9741):606-14. doi: 10.1016/S0140-6736(10)60889-6. Epub 2010 Aug 6. PMID 20692030

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 5 international sites - Ghana, Kenya, Mali, Bangladesh, and Vietnam from 29 March 2007 (first patient in) to 13 October 2008 (last dose given).
  Last subject completed follow-up: 31 March 2009
  All data corrections applied (Frozen File): 20 July 2009
Pre-assignment Details: Excluded from the trial before assignment to groups were subjects: with history of active gastrointestinal illness (vomiting, diarrhea, elevated temperature); who were participating in (or expected to participate in) other investigational-product studies; who could not be followed adequately for safety.
Groups:
- RotaTeq™ - Africa; RotaTeq™ - Asia: Three doses of RotaTeq™ (Rotavirus vaccine, live, oral, pentavalent) administered 28 to 70 days apart, with up to 14 days of safety follow-up after each vaccination, and follow-up for acute gastrointestinal episodes (AGEs) until the end of the study.
- Placebo - Africa; Placebo - Asia: Three doses of Placebo matching RotaTeq™ administered 28 to 70 days apart, with up to 14 days of safety follow-up after each vaccination and follow-up for acute gastrointestinal episodes (AGEs) until the end of the study.
Period: Overall Study
Arm/Group | RotaTeq™ - Africa | Placebo - Africa | RotaTeq™ - Asia | Placebo - Asia
Started | 2733 (Subjects who passed all entry criteria and who were randomized in to the study) | 2735 (Subjects who passed all entry criteria and who were randomized in to the study) | 1018 (Subjects who passed all entry criteria and who were randomized in to the study) | 1018 (Subjects who passed all entry criteria and who were randomized in to the study)
Vaccinated at Visit 1 | 2733 | 2735 | 1018 | 1018
Vaccinated at Visit 2 | 2657 | 2666 | 1013 | 1009
Vaccinated at Visit 3 | 2613 | 2612 | 1009 | 1007
Completed | 2607 (Subjects vaccinated and followed up to 14 days after each dose) | 2601 (Subjects vaccinated and followed up to 14 days after each dose) | 1009 (Subjects vaccinated and followed up to 14 days after each dose) | 1007 (Subjects vaccinated and followed up to 14 days after each dose)
Not Completed | 126 | 134 | 9 | 11
Not completed — Adverse Event | 12 | 21 | 1 | 0
Not completed — Lost to Follow-up | 62 | 69 | 4 | 3
Not completed — Protocol Violation | 4 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 48 | 42 | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RotaTeq™ - Africa | Placebo - Africa | RotaTeq™ - Asia | Placebo - Asia | Total
Number analyzed (Participants) | 2733 | 2735 | 1018 | 1018 | 7504
Age, Customized [Number; unit: participants]
  <27 Days | 0 | 1 | 0 | 0 | 1
  27 to 41 Days | 536 | 569 | 3 | 7 | 1115
  42 to 84 Days | 2197 | 2165 | 1015 | 1011 | 6388
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1359 | 1370 | 464 | 492 | 3685
  Male | 1374 | 1365 | 554 | 526 | 3819
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 2733 | 2735 | 0 | 0 | 5468
  Asian | 0 | 0 | 1017 | 1016 | 2033
  Multi-Racial | 0 | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Severe Clinical Rotavirus Disease Caused by Any Rotavirus Serotype More Than 14 Days Following the Third Dose
Time Frame: At least 14 days following the third vaccination
Population: Per Protocol Population
Measure: Number; unit: Subjects
Arm/Group | RotaTeq™ - Africa | Placebo - Africa | RotaTeq™ - Asia | Placebo - Asia
Number analyzed (Participants) | 2357 | 2348 | 991 | 978
Subjects
  Subjects with rotavirus gastroenteritis cases | 79 | 129 | 38 | 71
  Subjects without rotavirus gastroenteritis cases | 2278 | 2219 | 953 | 907
Statistical Analysis 1: Comparison: RotaTeq™ - Africa vs Placebo - Africa; The number randomized is different from the number analyzed because some data were excluded from the analysis: subjects were classified as unevaluable due to wildtype rotavirus in stool before 14 days Postdose 3, incomplete clinical and/or laboratory results, or stool samples collected out of day range. Rotavirus gastroenteritis cases are subjects with one or more positive episodes. The most severe positive episode is used for the date of the case; Test type: Superiority or Other; p < 0.001, Exact binomial test — Efficacy>0%. Based on p< 1/(1+k), where p is proportion of subjects with outcome in vaccine group relative to total number of subjects with outcome, and k is ratio of follow-up time; placebo / vaccine. Based on conditional binomial approach; Efficacy = 1-Relative Risk = 39.3, 95% CI [19.1 to 54.7] — Efficacy = 1-RR, expressed as a percentage; the RR is the incidence in the vaccine group / the incidence in the placebo group
Statistical Analysis 2: Comparison: RotaTeq™ - Asia vs Placebo - Asia; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Exact binomial test — [p-value comment as in outcome 1, analysis 1]; Efficacy = 1-Relative Risk = 48.3, 95% CI [22.3 to 66.1] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Africa - Serum Anti-rotavirus IgA Responses and Serum Neutralizing Antibody (SNA) Responses Against Rotavirus Serotypes G1, G2, G3, G4, and P1A[8]
Description: Induction of postdose 3 SNA response (Number of subjects with ≥ 3 fold rise in antibody titer)
Time Frame: 14 days following the 3rd vaccination
Population: Per Protocol Population
  *N analyzed for Serotype P1A[8] is 188
Measure: Number; unit: Subjects
Arm/Group | RotaTeq™ - Africa | Placebo - Africa
Number analyzed (Participants) | 189 | 169
Subjects
  ≥ 3 fold rise in anti-rotavirus IgA | 148 | 34
  ≥ 3 fold rise in antibody titer: Serotype G1 | 35 | 0
  ≥ 3 fold rise in antibody titer: Serotype G2 | 17 | 5
  ≥ 3 fold rise in antibody titer: Serotype G3 | 12 | 4
  ≥ 3 fold rise in antibody titer: Serotype G4 | 50 | 4
  ≥ 3 fold rise in antibody titer: Serotype P1A[8] | 27 | 8
Statistical Analysis 1: Comparison: RotaTeq™ - Africa; Anti-rotavirus IgA; Test type: Superiority or Other; Percentage = 78.3, 95% CI [71.7 to 84.0]
Statistical Analysis 2: Comparison: RotaTeq™ - Africa; Serotype G1; Test type: Superiority or Other; Percentage = 18.5, 95% CI [13.3 to 24.8]
Statistical Analysis 3: Comparison: RotaTeq™ - Africa; Serotype G2; Test type: Superiority or Other; Percentage = 9.0, 95% CI [5.3 to 14.0]
Statistical Analysis 4: Comparison: RotaTeq™ - Africa; Serotype G3; Test type: Superiority or Other; Percentage = 6.3, 95% CI [3.3 to 10.8]
Statistical Analysis 5: Comparison: RotaTeq™ - Africa; Serotype G4; Test type: Superiority or Other; Percentage = 26.5, 95% CI [20.3 to 33.3]
Statistical Analysis 6: Comparison: RotaTeq™ - Africa; Serotype P1A[8]; Test type: Superiority or Other; Percentage = 14.4, 95% CI [9.7 to 20.2]
Statistical Analysis 7: Comparison: Placebo - Africa; Anti-rotavirus IgA; Test type: Superiority or Other; Percentage = 20.1, 95% CI [14.4 to 27.0]
Statistical Analysis 8: Comparison: Placebo - Africa; Serotype G1; Test type: Superiority or Other; Percentage = 0.0, 95% CI [0.0 to 2.2]
Statistical Analysis 9: Comparison: Placebo - Africa; Serotype G2; Test type: Superiority or Other; Percentage = 3.0, 95% CI [1.0 to 6.8]
Statistical Analysis 10: Comparison: Placebo - Africa; Serotype G3; Test type: Superiority or Other; Percentage = 2.4, 95% CI [0.6 to 5.9]
Statistical Analysis 11: Comparison: Placebo - Africa; Serotype G4; Test type: Superiority or Other; Percentage = 2.4, 95% CI [0.6 to 5.9]
Statistical Analysis 12: Comparison: Placebo - Africa; Serotype P1A[8]; Test type: Superiority or Other; Percentage = 4.7, 95% CI [2.1 to 9.1]

3. Secondary Outcome: Asia - Serum Anti-rotavirus IgA Responses and Serum Neutralizing Antibody (SNA) Responses Against Rotavirus Serotypes G1, G2, G3, G4, and P1A[8]
Description: Induction of postdose 3 SNA response (Number of subjects with ≥ 3 fold rise in antibody titer)
Time Frame: 14 days following the 3rd vaccination
Population: Per Protocol Population
Measure: Number; unit: Subjects
Arm/Group | RotaTeq™ - Asia | Placebo - Asia
Number analyzed (Participants) | 131 | 132
Subjects
  ≥ 3 fold rise in anti-rotavirus IgA | 115 | 24
  ≥ 3 fold rise in antibody titer: Serotype G1 | 42 | 3
  ≥ 3 fold rise in antibody titer: Serotype G2 | 13 | 1
  ≥ 3 fold rise in antibody titer: Serotype G3 | 37 | 4
  ≥ 3 fold rise in antibody titer: Serotype G4 | 24 | 0
  ≥ 3 fold rise in antibody titer: Serotype P1A[8] | 36 | 7
Statistical Analysis 1: Comparison: RotaTeq™ - Asia; Anti-rotavirus IgA; Test type: Superiority or Other; Percentage = 87.8, 95% CI [80.9 to 92.9]
Statistical Analysis 2: Comparison: RotaTeq™ - Asia; Serotype G1; Test type: Superiority or Other; Percentage = 32.1, 95% CI [24.2 to 40.8]
Statistical Analysis 3: Comparison: RotaTeq™ - Asia; Serotype G2; Test type: Superiority or Other; Percentage = 9.9, 95% CI [5.4 to 16.4]
Statistical Analysis 4: Comparison: RotaTeq™ - Asia; Serotype G3; Test type: Superiority or Other; Percentage = 28.2, 95% CI [20.7 to 36.8]
Statistical Analysis 5: Comparison: RotaTeq™ - Asia; Serotype G4; Test type: Superiority or Other; Percentage = 18.3, 95% CI [12.1 to 26.0]
Statistical Analysis 6: Comparison: RotaTeq™ - Asia; Serotype P1A[8]; Test type: Superiority or Other; Percentage = 27.5, 95% CI [20.0 to 36.0]
Statistical Analysis 7: Comparison: Placebo - Asia; Anti-rotavirus IgA; Test type: Superiority or Other; Percentage = 18.2, 95% CI [12.0 to 25.8]
Statistical Analysis 8: Comparison: Placebo - Asia; Serotype G1; Test type: Superiority or Other; Percentage = 2.3, 95% CI [0.5 to 6.5]
Statistical Analysis 9: Comparison: Placebo - Asia; Serotype G2; Test type: Superiority or Other; Percentage = 0.8, 95% CI [0.0 to 4.1]
Statistical Analysis 10: Comparison: Placebo - Asia; Serotype G3; Test type: Superiority or Other; Percentage = 3.0, 95% CI [0.8 to 7.6]
Statistical Analysis 11: Comparison: Placebo - Asia; Serotype G4; Test type: Superiority or Other; Percentage = 0.0, 95% CI [0.0 to 2.8]
Statistical Analysis 12: Comparison: Placebo - Asia; Serotype P1A[8]; Test type: Superiority or Other; Percentage = 5.3, 95% CI [2.2 to 10.6]

ADVERSE EVENTS:
Time Frame: Serious clinical adverse experiences (SAE) were recorded for all randomized subjects for 14 days post any vaccination. Kenya Safety Cohort subjects were followed for all nonserious and serious adverse experiences for 42 days post any vaccination.
Description: For SAFETY displays (SAEs and Other Adverse Events); SAE information is reported by treatment received and not reported by Region or subset. Other Adverse Events were only recorded for a subset of subjects (Kenya Safety Cohort, N=301), who were followed for all Other Adverse Events and SAEs occurring within 42 days following any vaccination.
Groups:
- RotaTeq™: Three doses of RotaTeq™ (Rotavirus vaccine, live, oral, pentavalent) administered 28 to 70 days apart, with up to 14 days of safety follow-up after each vaccination, and follow-up for acute gastrointestinal episodes (AGEs) until the end of the study.
  Serious clinical adverse experiences (SAE) were recorded for all randomized subjects for 14 days following any vaccination and are reported by treatment group (including cross treated subjects) and are not reported by Region (Africa and Asia).
  Other Adverse Events were recorded for a subset of subjects (Kenya Safety Cohort, N=301), who were followed for all non-serious and serious adverse experiences occurring within 42 days following any vaccination.
- Placebo: Three doses of Placebo matching RotaTeq™ administered 28 to 70 days apart, with up to 14 days of safety follow-up after each vaccination and follow-up for acute gastrointestinal episodes (AGEs) until the end of the study.
  SAEs were recorded for all randomized subjects for 14 days following any vaccination and are reported by treatment group (including cross treated subjects) and are not reported by Region (Africa and Asia).
  Other Adverse Events were recorded for a subset of subjects (Kenya Safety Cohort, N=301), who were followed for all non-serious and serious adverse experiences occurring within 42 days following any vaccination.
- RotaTeq™, Placebo, RotaTeq™; Placebo, Placebo, RotaTeq™: Includes SAE data for subjects who were cross-treated, ie; received a treatment other than what they were assigned.
  Serious clinical adverse experiences (SAE) were recorded for all randomized subjects for 14 days following any vaccination.
- RotaTeq™ - Kenya Safety Cohort; Placebo - Kenya Safety Cohort: A subset of subjects (Kenya Safety Cohort, N=301), were followed for all Other Adverse Events and SAEs occurring within 42 days following any vaccination.
Arm/Group | RotaTeq™ | Placebo | RotaTeq™, Placebo, RotaTeq™ | Placebo, Placebo, RotaTeq™ | RotaTeq™ - Kenya Safety Cohort | Placebo - Kenya Safety Cohort
Serious Adverse Events (participants affected / at risk) | 144/3744 | 156/3745 | 1/3 | 0/1 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 137/149 | 147/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RotaTeq™ (N=3744) | Placebo (N=3745) | RotaTeq™, Placebo, RotaTeq™ (N=3) | Placebo, Placebo, RotaTeq™ (N=1) | RotaTeq™ - Kenya Safety Cohort (N=0) | Placebo - Kenya Safety Cohort (N=0)
Anemia (Blood and lymphatic system disorders) | 8 | 5 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 4 | 0 | 0 | 0 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Vietnam had 1 confirmed case of intussusception (placebo recipient) subject was treated & fully recovered. The reporting investigator determined the serious event of clinical interest, was of moderate intensity, & not related to the study vaccine.
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 5 | 7 | 0 | 0 | 0 | 0
Drowning (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 1 | 0 | 0 | 0 | 0
Sudden infant death syndrome (General disorders) | 1 | 2 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 4 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 6 | 9 | 0 | 0 | 0 | 0
Cerebral malaria (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Dysentery (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Febrile infection (Infections and infestations) | 2 | 4 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 44 | 49 | 0 | 0 | 0 | 0
HIV infection (Infections and infestations) | 6 | 7 | 0 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Malaria (Infections and infestations) | 34 | 32 | 0 | 0 | 0 | 0
Meningitis (Infections and infestations) | 4 | 6 | 0 | 0 | 0 | 0
Meningitis pneumococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Omphalitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Oral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 46 | 44 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 7 | 9 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Salmonellosis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 4 | 0 | 0 | 0 | 0
Tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Typhoid fever (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Chemical poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Snake bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 3 | 3 | 0 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0
Feeding disorder of infancy or early childhood (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 5 | 4 | 0 | 0 | 0 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hepatoblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RotaTeq™ (N=0) | Placebo (N=0) | RotaTeq™, Placebo, RotaTeq™ (N=0) | Placebo, Placebo, RotaTeq™ (N=0) | RotaTeq™ - Kenya Safety Cohort (N=149) | Placebo - Kenya Safety Cohort (N=152)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 4
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 10 | 13
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 3
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 71 | 67
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 2
Faeces hard (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 35 | 31
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 2 | 2
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 96 | 98
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Abscess of eyelid (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 5 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 10 | 8
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Dysentery (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 39 | 45
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Malaria (Infections and infestations) | 0 | 0 | 0 | 0 | 23 | 34
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 3
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 15 | 14
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 16 | 19
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 4
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 54 | 62
Septic rash (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 3
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Tinea capitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 4
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Umbilical sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 5 | 6
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Tongue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Feeding disorder of infancy or early childhood (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Crying (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Fontanelle bulging (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 7 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 89 | 90
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 22 | 23
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 30 | 18
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 5 | 8
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pemphigus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pityriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 57 | 56
Rash generalized (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.